CLINICAL TRIAL: NCT01153880
Title: Pharmacovigilence for Retapamulin: Age-stratified Monitoring of Prescribed Use in the United States
Brief Title: United States Pharmacovigilence Retapamulin-Prescribing
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113158
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2013-05

CONDITIONS: Skin Infections, Bacterial
Keywords: Altabax; United States; topical; Mupirocin; Retapamulin; Bactroban
MeSH Terms: conditions — Cellulitis | interventions — retapamulin; Mupirocin

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Age <9 months definitive: Age at time of prescription was <9 months
  Interventions: Drug: Retapamulin; Drug: Co-prescription of retapamulin and topical mupirocin
- Age <9 months uncertain: Age at time of prescription was uncertain for <9 months
  Interventions: Drug: Retapamulin; Drug: Co-prescription of retapamulin and topical mupirocin
- 9 months to 6 years: Age at time of prescription was 9 months to 6 years
  Interventions: Drug: Retapamulin; Drug: Co-prescription of retapamulin and topical mupirocin
- 7 to 18 years: Age at time of prescription was 7 to 18 years
  Interventions: Drug: Retapamulin; Drug: Co-prescription of retapamulin and topical mupirocin
- 19 to 65 years: Age at time of prescription was 19 to 65 years
  Interventions: Drug: Retapamulin; Drug: Co-prescription of retapamulin and topical mupirocin
- 66 years and older: Age at time of prescription was 66 years and older
  Interventions: Drug: Retapamulin; Drug: Co-prescription of retapamulin and topical mupirocin

INTERVENTIONS:
Drug: Retapamulin — Prescription sales claim of retapamulin
Drug: Co-prescription of retapamulin and topical mupirocin — Same day prescription sales claims for retapamulin and topical mupirocin

SUMMARY:
Retapamulin, a topical pleuromutilin antibiotic, is the first in a new class of topical antibiotics approved for human use. In the United States (US), retapamulin is approved for the treatment of impetigo in persons nine or more months of age and was launched on 12 April 2007. This five-year study is designed to examine use of retapamulin in the pediatric population less than nine months of age. We will conduct an annual assessment of prescription sales claims for retapamulin using the Integrated Health Care Information Services (IHCIS) National Managed Care Benchmarked Database. For each year of reporting, the observed frequencies of the exposure, with or without same-day, co-prescribed sales claim of mupirocin, will be identified. The study objectives are to determine the frequency of retapamulin sales in a representative US population stratified by the designated age group and to determine the frequency of same-day sale of the topical agent, mupirocin.

DETAILED DESCRIPTION:
The IHCIS is Health Insurance Portability and Accountability Act (HIPAA) compliant with encrypted member and provider identifiers; date of birth is restricted to year of birth. Based on year of birth and the prescription sales claim date, age at the time of the prescription(s) will be categorized as less than 9 months (definitive) and less than 9 months (uncertain).

ELIGIBILITY:
Inclusion Criteria:

* The study population will consist of all 'eligible members' in the IHCIS database with a valid gender and age record who have at least 1 month enrolment and eligibility of pharmacy benefits.

Exclusion Criteria:

* Membership in IHCIS without a valid gender or age record, enrolment less than 1 month, or ineligibility for pharmacy benefits will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Members with enrollment and phamacy benefits eligibility in the Integrated Health Care Information Services (IHCIS) National Managed Care Benchmarked Database will be assessed annually for prescription sales claims for five years post-launch of retapamulin. The IHCIS is a US national managed care database which is Health Insurance Portability and Accountability Act (HIPAA) compliant and features encrypted member and provider identifiers.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2008-12; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Prescription of retapamulin | First prescription in database for each calendar year between January 2007 and December 2011

SECONDARY OUTCOMES:
Prescription for retapamulin and topical mupirocin | First same-day prescriptions for both medicines in database for each calendar year between Janaury 2007 and December 2011

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline